CLINICAL TRIAL: NCT04403347
Title: Effect of Tartary Buckwheat Diet Intervention on Primary Hypertension and the Underlying Mechanism of Gut Microbiome Restoration
Brief Title: Effect of Gut Microbiome Restoration on Primary Hypertension Via Dietary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Director, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-GZ10 (Part II)
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: Hypertension; Microbiome; Treatment; Diet
MeSH Terms: conditions — Hypertension | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative Dietary Formulation (Experimental): In addition to adherence to a regular diet and usual hypertension care, participants will receive an innovative dietary formulation (TBW diet) incorporated into their daily meals and administered orally.
  Interventions: Dietary Supplement: Innovative Dietary Formulation (Patent ID: CN110250417A)
- Usual Care (Other): Usual Care (Guideline-based patient education and lifestyle recommendations)
  Interventions: Other: Regular Diet

INTERVENTIONS:
Dietary Supplement: Innovative Dietary Formulation (Patent ID: CN110250417A) — In addition to adherence to a regular diet and standard hypertension care, participants will receive an innovative dietary formulation incorporated into their daily meals and administered orally.
  Arms: Innovative Dietary Formulation
Other: Regular Diet — Regular Diet with Usual Care
  Arms: Usual Care

SUMMARY:
Mounting preclinical and clinical evidences have proved the optimal role of diets (i.e. DASH (Dietary Approaches to Stop Hypertension) diet, Mediterranean diet) on BP control and a causal role of gut microbiota on the pathogenesis of primary hypertension. Dietary changes appeared to reshape gut microbiota and to ameliorate diseases such as Type 2 Diabetes. A hypothesis is thus raised that dietary changes can be a potential approach to ameliorate hypertension via gut microbiome restoration. This pilot study will utilize an innovative natural dietary formulation (patent ID: CN110250417A) derived from Tartary buckwheat(TBW) diet, in comparison with usual care (guideline-based patient education and lifestyle recommendations), to investigate its effect and safety on primary hypertension treatment, and the underlying mechanisms of gut microbiome restoration.

DETAILED DESCRIPTION:
Primary hypertension is a most prevalent cardiovascular diseases, and becomes a severe global public health issue because of the high morbidity and potential risk to other cardiovascular diseases. Several animal studies and diverse patient cohorts reported that the disorder of gut microbiome correlated with hypertension. Based on the investigators' previous work findings of metagenomics analysis, fecal transplantation and metabolomics changes in hypertension and pre-hypertension patients, a casual role of gut microbiome disorder was observed in primary hypertension and raised a hypothesis that gut microbiome restoration can be a potential approach to ameliorate hypertension. Recent studies indicated FMT, prebiotics, probiotics, dietary changes and other methodologies can assist gut microbiome restoration in diseases such as type 2 diabetes. The investigators therefore develop two pilot studies respectively utilizing FMT capsules (Pilot Study I) and innovative dietary changes (Pilot Study II) to explore the methodologies, effect, safety and underlying mechanisms of gut microbiome restoration on hypertension. These pilot studies also present as the clinical translational part of the research project "The Role of Gut Microbiome in the Pathogenesis of Essential Hypertension"(Project ID 81630014, sponsored by National Natural Science Foundation of China).

This study is the Pilot Study II:

Objective: With reference of DASH diet and Mediterranean diet, this study aims to explore the effect and safety of an innovative natural dietary formulation (deriving from TBW diet) on primary hypertension, and the underlying mechanisms of gut microbiome restoration.

Study Design: A multicenter, randomized, open-label, controlled study.

Data quality control and statistical analysis: The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality.

Ethics: The Ethics Committee of Fuwai Hospital approved this study. Informed consents before patient enrollment are required.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~60 years.
2. Established Diagnosis of Grade 1 Hypertension (initial diagnosis or free from antihypertensive drugs within a month): 140mmHg≤ Office SBP<160mmHg for three measurements at different days without any antihypertensive medications, according to the "2010 Chinese Guidelines for Prevention and Treatment of Hypertension".
3. Patients with informed consent after thorough explanation.

Exclusion Criteria:

1. Antibiotics or probiotics usage within last 4 weeks
2. Participants of other clinical trials related to hypertension currently or within last 3 months
3. Antihypertensive medications usage currently or within last month
4. Diagnosed secondary hypertension
5. Severe hepatic or renal diseases ((ALT >3 times the upper limit of normal value, or end stage renal disease on dialysis or eGFR <30 mL/min/1.73 m2, or serum creatinine >2.5 mg/dl [>221 μmol/L])
6. History of large atherosclerotic cerebral infarction or hemorrhagic stroke (not including lacunar infarction and transient ischemic attack [TIA])
7. Hospitalization for myocardial infarction within last 6 months; Coronary revascularization (PCI or CABG) within last 12 months; Planned for PCI or CABG in the next 12 months.
8. Sustained atrial fibrillation or arrhythmias at recruitment disturbing the electronic BP measurement.
9. NYHA class III-IV heart failure; Hospitalization for chronic heart failure exacerbation within last 6 months.
10. Severe valvular diseases; Potential for surgery or percutaneous valve replacement within the study period.
11. Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Rheumatic heart disease; Congenital heart disease.
12. Other severe diseases influencing the entry or survival of participants, such as malignant tumor or acquired immune deficiency syndrome.
13. Cognitive impairment or severe neuropsychiatric comorbidities who are incapable of providing their own informed consent.
14. Participants preparing for or under pregnancy and/or lactation.
15. Other conditions inappropriate for recruitment according to the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Change for Office Systolic Blood Pressure (SBP) | From Baseline to the Month 2 (Week 8) follow-up visit
  Change for Office Systolic Blood Pressure (SBP)

SECONDARY OUTCOMES:
Change for office SBP | Baseline, Month 1(Week 4), Month 3(Week 12)
  Change for office SBP
Change for Office Diastolic Blood Pressure (DBP) | Baseline, Month 1(Week 4), Month 2 (Week 8), Month 3 (Week 12)
  Change for Office Diastolic Blood Pressure (DBP)
Change for daytime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Change for daytime average SBP via 24-hour Ambulatory BP Monitoring
Change for daytime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Change for daytime average DBP via 24-hour Ambulatory BP Monitoring
Change for nighttime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Change for nighttime average SBP via 24-hour Ambulatory BP Monitoring
Change for nighttime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Change for nighttime average DBP via 24-hour Ambulatory BP Monitoring
Number of Participants with Adverse Events (AEs) as a Measure of Safety | All AEs over 3 months
  Number of Participants with Adverse Events (AEs) as a Measure of Safety
Intestinal Microbiota Composition Pre- and Post-intervention (innovative dietary formulation or usual care) via Metagenomic Analysis | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Intestinal Microbiota Composition Pre- and Post-intervention (innovative dietary formulation or usual care) via Metagenomic Analysis
Intestinal Microbiota function Pre- and Post-intervention (innovative dietary formulation or usual care) via Metagenomic Analysis | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Intestinal Microbiota function Pre- and Post-intervention (innovative dietary formulation or usual care) via Metagenomic Analysis
Plasma Metabolite Composition Pre- and Post-intervention (innovative dietary formulation or usual care) via Metabolomic Analysis | Baseline, Month 1(Week 4), Month 2(Week 8), Month 3(Week 12)
  Plasma Metabolite Composition Pre- and Post-intervention (innovative dietary formulation or usual care) via Metabolomic Analysis
Change for Fasting Blood Glucose Level | Baseline, Month 2(Week 8)
  Change for Fasting Blood Glucose Level
Change for Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol) | Baseline, Month 2(Week 8)
  Change for Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol)
Change for Body Mass Index | Baseline, Month 2(Week 8)
  Change for Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD,PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (8):
- China (8):
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Clinical Medical College&Affiliated Hospital of Chengdu University, Chengdu, Sichuan
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - the People's Hospital of Ji Xian District, Tianjin

REFERENCES:
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Zhao L, Zhang F, Ding X, Wu G, Lam YY, Wang X, Fu H, Xue X, Lu C, Ma J, Yu L, Xu C, Ren Z, Xu Y, Xu S, Shen H, Zhu X, Shi Y, Shen Q, Dong W, Liu R, Ling Y, Zeng Y, Wang X, Zhang Q, Wang J, Wang L, Wu Y, Zeng B, Wei H, Zhang M, Peng Y, Zhang C. Gut bacteria selectively promoted by dietary fibers alleviate type 2 diabetes. Science. 2018 Mar 9;359(6380):1151-1156. doi: 10.1126/science.aao5774. PMID 29590046
- [Background] Marques FZ, Nelson E, Chu PY, Horlock D, Fiedler A, Ziemann M, Tan JK, Kuruppu S, Rajapakse NW, El-Osta A, Mackay CR, Kaye DM. High-Fiber Diet and Acetate Supplementation Change the Gut Microbiota and Prevent the Development of Hypertension and Heart Failure in Hypertensive Mice. Circulation. 2017 Mar 7;135(10):964-977. doi: 10.1161/CIRCULATIONAHA.116.024545. Epub 2016 Dec 7. PMID 27927713